CLINICAL TRIAL: NCT03371017
Title: A Phase III, Randomised, Double-Blind, Placebo-Controlled, Multicentre Study Of The Efficacy And Safety Of Atezolizumab Plus Chemotherapy For Patients With Early Relapsing Recurrent (Inoperable Locally Advanced Or Metastatic) Triple-Negative Breast Cancer
Brief Title: A Study of the Efficacy and Safety of Atezolizumab Plus Chemotherapy for Patients With Early Relapsing Recurrent Triple-Negative Breast Cancer
Acronym: IMpassion132
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MO39193; 2016-005119-42 (EudraCT Number)
Record Dates: First submitted 2017-11-21; First posted 2017-12-13 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Triple Negative Breast Neoplasms
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; Gemcitabine; Capecitabine; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab (Experimental): Participants will receive Atezolizumab on day 1 of each 3-week treatment cycle
  Interventions: Drug: Atezolizumab; Drug: Gemcitabine; Drug: Capecitabine; Drug: Carboplatin
- Placebo (Placebo Comparator): Participants will receive Placebo on day 1 of each 3-week treatment cycle
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Capecitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered, 1200 mg by IV infusion with :
  gemcitabine 1000 mg/m2, followed by carboplatin target area under the curve (AUC) 2 mg/ml/min, both administered by IV infusion on Days 1 and 8 of each 3-week treatment cycle or with capecitabine 1000 mg/m2, twice daily orally on Days 1 to 14, followed by a 7-day rest period in each 3-week treatment cycle
  Arms: Atezolizumab
Drug: Placebo — Placebo will be administered, 1200 mg by IV infusion with :
  gemcitabine 1000 mg/m2, followed by carboplatin target area under the curve (AUC) 2 mg/ml/min, both administered by IV infusion on Days 1 and 8 of each 3-week treatment cycle or with capecitabine 1000 mg/m2, twice daily orally on Days 1 to 14, followed by a 7-day rest period in each 3-week treatment cycle
  Arms: Placebo
Drug: Gemcitabine — Gemcitabine 1000 mg/m2, followed by carboplatin target area under the curve (AUC) 2 mg/ml/min, both administered by IV infusion on Days 1 and 8 of each 3-week treatment cycle
Drug: Capecitabine — Capecitabine 1000 mg/m2, twice daily orally on Days 1 to 14, followed by a 7-day rest period in each 3-week treatment cycle
Drug: Carboplatin — Carboplatin target area under the curve (AUC) 2 mg/ml/min, both administered by IV infusion on Days 1 and 8 of each 3-week treatment cycle

SUMMARY:
This study will evaluate the efficacy and safety of atezolizumab plus chemotherapy compared with placebo plus chemotherapy in patients with inoperable recurrent triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed triple negative breast cancer (TNBC) that is either locally recurrent, inoperable and cannot be treated with curative intent or is metastatic
* Documented disease progression occurring within 12 months from the last treatment with curative intent
* Prior treatment (of early breast cancer) with an anthracycline and taxane
* Have not received prior chemotherapy or targeted systemic therapy for their locally advanced inoperable or metastatic recurrence. Prior radiation therapy for recurrent disease is permitted
* Measurable or non-measurable disease, as defined by RECIST 1.1
* Availability of a representative formalin-fixed, paraffin-embedded (FFPE) tumour block (preferred) or at least 17 unstained slides obtained from relapsed metastatic or locally advanced diseases may be submitted, if clinically feasible, with an associated pathology report, if available. If a fresh tumour sample is not clinically feasible, either the diagnosis sample, the primary surgical resection sample, or the most recent FFPE tumour biopsy sample should be used.
* Eastern Cooperative Oncology Group performance status 0-1
* Life expectancy ≥ 12 weeks
* Adequate haematologic and end-organ function
* Negative human immunodeficiency virus (HIV) test ---Negative hepatitis B surface antigen (HBsAg) test at screening
* Negative total hepatitis B core antibody (HBcAb) test at screening, or positive HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening
* The HBV DNA test will be performed only for patients who have a negative HBsAg and a positive HBcAb test.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening.
* Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of ≤1% per year during the treatment period and for at least 5 months after the last dose of atezolizumab or 6 months after the last dose of capecitabine, whichever is later. In addition, women must refrain from donating eggs during the same time period.
* Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm

Inclusion criteria for patients enrolled after the recruitment of all-comers is complete:

-PD-L1-positive tumour status (assessed centrally prior to randomisation), defined as PD-L1 expression on tumour-infiltrating immune cells (IC) of 1% or greater.

Exclusion Criteria:

* Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to randomisation
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.
* Symptomatic or rapid visceral progression
* No prior treatment with an anthracycline and taxane
* History of leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) (patients with indwelling catheters such as PleurX® are allowed)
* Uncontrolled tumour-related pain
* Uncontrolled or symptomatic hypercalcemia
* Malignancies other than TNBC within 5 years prior to randomisation)
* Significant cardiovascular disease, within 3 months prior to randomisation, unstable arrhythmias, or unstable angina
* Presence of an abnormal ECG
* Severe infection requiring oral or IV antibiotics within 4 weeks prior to randomisation, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
* Current treatment with anti-viral therapy for HBV.
* Major surgical procedure within 4 weeks prior to randomisation or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis
* Treatment with investigational therapy within 28 days prior to randomisation
* Pregnant or lactating, or intending to become pregnant during or within 5 months after the last dose of atezolizumab, or within 6 months after the last dose of capecitabine, whichever is later.

Exclusion Criteria Related to Atezolizumab:

* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanised antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or to any component of the atezolizumab formulation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computerised tomography (CT) scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active tuberculosis
* Receipt of a live, attenuated vaccine within 4 weeks prior to randomisation or anticipation that a live, attenuated vaccine will be required during atezolizumab/placebo treatment or within 5 months after the last dose of atezolizumab/placebo
* Prior treatment with CD137 agonists, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin [IL]-2) within 4 weeks or five half-lives of the drug (whichever is longer) prior to randomisation
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to start of study treatment, or anticipated requirement for systemic immunosuppressive medications during the trial

Exclusion Criteria Related to Capecitabine:

* Inability to swallow pills
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, or ulcerative colitis
* Known dihydropyrimidine dehydrogenase (DPD) deficiency or history of severe and unexpected reactions to fluoropyrimidine therapy in patients selected to receive capecitabine

Exclusion Criteria Related to Carboplatin/Gemcitabine:

-Hypersensitivity to platinum containing compounds or any component of carboplatin or gemcitabine drug formulations in patients selected to receive carboplatin and Gemcitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (124):
- United States (6):
  - Florida Cancer Specialists - Fort Myers (Broadway), Fort Myers, Florida
  - Florida Cancer Specialists & Research Institute, St. Petersburg, Florida
  - The Valley Hospital, Paramus, New Jersey
  - Magee-Woman's Hospital, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Argentina (2):
  - Hospital Provincial del Centenario, Rosario
  - Instituto de Oncología de Rosario, Rosario
- Clinical center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (9):
  - Oncocentro Serviços Medicos E Hospitalares Ltda, Fortaleza, Ceará
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Centro de Oncologia de Santa Catarina LTDA, Chapecó, Santa Catarina
  - Instituto de Pesquisa Grupo NotreDame Intermedica, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo, São Paulo
- Chile (2):
  - Bradford Hill Centro de Investigaciones Clinicas, Recoleta
  - Clinica Vespucio, Santiago
- China (18):
  - the First Affiliated Hospital of Bengbu Medical College, Anhui
  - Cancer Hospital , Chinese Academy of Medical, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fujian
  - Sun Yat-sen Memorial Hospital, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital Of Jinzhou Medical University, Jinzhou
  - Jiangsu Province Hospital, Nanjing
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanxi Province Cancer Hospital, Taiyuan
  - Tianjin Cancer Hospital, Tianjin
  - The First Affiliated Hospital of The Fourth Military Medical University (Xijing Hospital), Xi'an
- Cuba (2):
  - Hospital Hermanos Ameijeiras, La Habana
  - Instituto Nacional de Oncología y Radiología (INOR), La Habana
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- France (7):
  - Centre Georges-François Lecler, Dijon
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Régional de Lutte Contre Le Cancer Val D'aurelle Paul Lamarque, Montpellier
  - Centre Eugene Marquis, Rennes
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - IGR, Villejuif
- Germany (7):
  - Universitätsklinikum "Carl Gustav Carus", Dresden
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH, Essen
  - Varisano Klinikum Frankfurt Höchst GmbH, Frankfurt
  - Universitätsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover, Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Medizinisches Zentrum für Hämatologie und Onkologie, München
- Hungary (5):
  - Szent Margit Hospital, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Pécsi Tudományegyetem, Pécs
- Italy (9):
  - Ospedale Antonio Perrino, Brindisi, Apulia
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliero Universitaria San Martino, Genoa, Liguria
  - Ospedale San Raffaele S.r.l., Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo, Candiolo, Piedmont
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Kazakh Scientific Research Institution Of Oncology and Radiology, Almaty, Kazakhstan
- Mexico (3):
  - Centro Medico Dalinde, Mexico City, Mexico CITY (federal District)
  - Instituto Nacional de Cancerologia, Distrito Federal
  - CENEIT Oncologicos, Mexico City
- Clinical Center of Montenegro, Podgorica, Montenegro
- Morocco (3):
  - Centre Hospitalier Universitaire Hassan II, Fes
  - Centre Hospitalier Universitaire Mohamed VI, Marrakesh
  - Clinique specialise Menara, Marrakesh
- The Panama Clinic, Panama City, Panama
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Poland (2):
  - ?wi?tokrzyskie Centrum Onkologii, Kielce
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad, Warsaw
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto ? Hospital de Santo António, Porto
- Russia (6):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - Moscow Clinical Scientific Center, Moscow, Moscow Oblast
  - FSBI "National Medical Research Center of Oncology N.N. Blokhin?, Moscow, Moscow Oblast
  - Private Healthcare Institution Clinical Hospital RZhD Medicine, Saint Petersburg, Sankt-Peterburg
  - City Clinical Oncology Dispensary, SPb SBIH CCOD, Saint Petersburg, Sankt-Peterburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg, Sankt-Peterburg
- Serbia (4):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Clinical Centre Nis, Clinic for Oncology, Niš
- National Cancer Centre, Singapore, Singapore
- South Africa (3):
  - Wits Clinical Research, Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Private Oncology Centre, Pretoria
- South Korea (5):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital de Cruces, Bilbao, Vizcaya
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia
- Turkey (Türkiye) (6):
  - Ankara Oncology Hospital, Ankara
  - Ege University Medical Faculty, Bornova, ?zm?r
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Medipol University Medical Faculty, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Necmettin Erbakan University Meram Medical Faculty, Konya
- United Kingdom (9):
  - Velindre Cancer Centre, Cardiff
  - University Hospital Coventry, Coventry
  - Western General Hospital, Edinburgh
  - Royal Lancaster Infirmary, Morecambe Bay Hospitals Nhs Trust, Lancaster
  - Barts, London
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Mount Vernon Cancer Centre, Northwood
  - Royal Stoke University Hospital, Stoke-on-Trent

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 595 participants with inoperable locally advanced or metastatic Triple-negative Breast Cancer (TNBC) took part in the study at 126 investigative sites in 28 countries from 11 January 2018 to 23 October 2024.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive atezolizumab with chemotherapy or placebo with chemotherapy.
Groups:
- Placebo + Chemotherapy: Participants received atezolizumab matching placebo by intravenous (IV) infusion on Day 1 of each cycle along with either gemcitabine, 1000 milligrams per square meter (mg/m^2), followed by carboplatin target under the curve (AUC) 2 milligrams per milliliter per minute (mg/ml/min), both administered by IV infusion on Days 1 and 8 of each cycle or capecitabine, 1000 mg/m^2, twice daily (BID), orally on Days 1 to 14, followed by a 7-day rest period in each cycle (1 Cycle= 3 weeks). Treatment was continued until disease progression (PD), unacceptable toxicity, death or participant or investigator decision to discontinue treatment.
- Atezolizumab + Chemotherapy: Participants received atezolizumab 1200 milligrams (mg), by IV infusion on Day 1 of each cycle along with either gemcitabine, 1000 mg/m^2, followed by carboplatin target AUC 2 mg/ml/min, both administered by IV infusion on Days 1 and 8 of each cycle or capecitabine, 1000 mg/m^2, BID, orally on Days 1 to 14, followed by a 7-day rest period in each cycle (1 Cycle = 3 weeks). Treatment was continued until PD, unacceptable toxicity, death or participant or investigator decision to discontinue treatment.
Period: Overall Study
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Started | 298 | 297
Safety-evaluable Population (Safety-evaluable population included participants who received any amount of any study drug (atezolizumab/placebo or chemotherapy).) | 294 | 293
Programmed Death-ligand 1 (PD-L1)-Positive Population (PD-L1 positive population included all participants randomized in the study whose PD-L1 status was tumor-infiltrating immune cells (IC) of 1% or greater (IC1/2/3) at the time of randomization, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received.) | 177 | 177
Modified Intent-to-Treat (mITT) Population (mITT population included all participants randomized under the protocol versions prior to version 4.0 (referred to as all-comers, i.e., PD-L1(SP142)-positive and PD-L1(SP142)-negative participants), grouped according to their assigned treatment arm, whether or not the assigned study treatment was received.) | 192 | 188
Completed | 0 | 0
Not Completed | 298 | 297
Not completed — Physician Decision | 0 | 1
Not completed — Reason not Specified | 0 | 1
Not completed — Lost to Follow-up | 13 | 16
Not completed — Death | 228 | 215
Not completed — Withdrawal by Subject | 20 | 25
Not completed — Study Ended by Sponsor | 37 | 38
Not completed — Protocol Deviation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all participants randomized in the study, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received.
Groups:
- Placebo + Chemotherapy: Participants received atezolizumab matching placebo, by IV infusion on Day 1 of each cycle along with either gemcitabine, 1000 mg/m^2, followed by carboplatin target AUC 2 mg/ml/min, both administered by IV infusion on Days 1 and 8 of each cycle or capecitabine, 1000 mg/m^2, BID, orally on Days 1 to 14, followed by a 7-day rest period in each cycle (1 Cycle= 3 weeks). Treatment was continued until PD, unacceptable toxicity, death or participant or investigator decision to discontinue treatment.
- Atezolizumab + Chemotherapy: Participants received atezolizumab 1200 mg, by IV infusion on Day 1 of each cycle along with either gemcitabine, 1000 mg/m^2, followed by carboplatin target AUC 2 mg/ml/min, both administered by IV infusion on Days 1 and 8 of each cycle or capecitabine, 1000 mg/m^2, BID, orally on Days 1 to 14, followed by a 7-day rest period in each cycle (1 Cycle = 3 weeks). Treatment was continued until PD, unacceptable toxicity, death or participant or investigator decision to discontinue treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy | Total
Number analyzed (Participants) | 298 | 297 | 595
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.7) | 48.6 (10.9) | 49.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 297 | 595
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 51 | 110
  Not Hispanic or Latino | 222 | 218 | 440
  Unknown or Not Reported | 17 | 28 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 5 | 8
  Asian | 66 | 69 | 135
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 199 | 184 | 383
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 20 | 28 | 48

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in PD-L1-positive Population
Description: OS was defined as time from randomization to death from any cause. Participants without a reported death event at the time of the analysis were censored on the date they were last known to be alive. If no post-baseline data were available, OS was censored at the date of randomization +1 day.
Time Frame: Time from randomization to death (Up to 68 months)
Population: PD-L1 positive population included all participants randomized in the study whose PD-L1 status was tumor-infiltrating IC of 1% or greater (IC1/2/3) at the time of randomization, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 177 | 177
months | 11.24 [9.00 to 13.31] | 12.09 [10.12 to 15.08]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.5891, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.73 to 1.20]

2. Primary Outcome: OS in Modified Intent-to-treat (mITT) Population
Description: as for outcome 1
Time Frame: Time from randomization to death (Up to 68 months)
Population: mITT population included all participants randomized under the protocol versions prior to version 4.0 (referred to as all-comers, i.e., PD-L1(SP142)-positive and PD-L1(SP142)-negative participants, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 192 | 188
months | 9.79 [8.44 to 11.96] | 10.35 [8.90 to 12.88]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.6139, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.76 to 1.18]

3. Secondary Outcome: 12-month Survival Rate in PD-L1-positive Population
Description: 12-month survival rate was defined as the percentage of participants alive 12 months after randomization. The 12-month survival rates were estimated by Kaplan-Meier methodology. Percentages have been rounded off to the nearest whole number.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 177 | 177
percentage of participants | 47.58 [39.92 to 55.23] | 50.26 [42.61 to 57.91]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.6264, Z-test; Difference in Event Free Rate = 2.69, 95% CI 2-sided [-8.14 to 13.51]

4. Secondary Outcome: 12-month Survival Rate in mITT Population
Description: 12-month survival rate was defined as the percentage of participants alive 12 months after randomization. The 12-month survival rates were estimated by Kaplan-Meier methodology. Percentages have been rounded off to nearest whole number.
Time Frame: 12 months
Population: mITT population included all participants randomized under the protocol versions prior to version 4.0 (referred to as all-comers, i.e., PD-L1(SP142)-positive and PD-L1(SP142)-negative participants), grouped according to their assigned treatment arm, whether or not the assigned study treatment was received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 192 | 188
percentage of participants | 42.44 [35.23 to 49.66] | 46.20 [38.84 to 53.56]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.4750, Z-test; Difference in Event Free Rate = 3.76, 95% CI 2-sided [-6.55 to 14.07]

5. Secondary Outcome: 18-month Survival Rate in PD-L1-positive Population
Description: 18-month survival rate was defined as the percentage of participants alive 18 months after randomization. The 18-month survival rates were estimated by Kaplan-Meier methodology. Percentages have been rounded off to nearest whole number.
Time Frame: 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 177 | 177
percentage of participants | 32.48 [25.07 to 39.89] | 33.63 [26.05 to 41.21]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.8315, Z-test; Difference in Event Free Rate = 1.15, 95% CI 2-sided [-9.45 to 11.75]

6. Secondary Outcome: 18-month Survival Rate in mITT Population
Description: as for outcome 5
Time Frame: 18 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 192 | 188
percentage of participants | 25.68 [19.15 to 32.21] | 27.05 [20.39 to 33.71]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.7738, Z-test; Difference in Event Free Rate = 1.37, 95% CI 2-sided [-7.96 to 10.69]

7. Secondary Outcome: Progression-free Survival (PFS) in PD-L1-positive Population
Description: PFS was defined as the time from randomization to the first occurrence of PD, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1), or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 millimeters (mm). Data for participants not experiencing PD or death were censored at the last tumour assessment date. If no tumor assessment was performed after randomisation, data were censored at the date of randomisation +1 day.
Time Frame: Time from randomization to the first occurrence of PD or death (Up to 68 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 177 | 177
months | 3.58 [3.35 to 4.17] | 4.21 [3.71 to 5.62]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.1387, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.06]

8. Secondary Outcome: PFS in mITT Population
Description: PFS was defined as the time from randomization to the first occurrence of PD, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Data for participants not experiencing PD or death were censored at the last tumour assessment date. If no tumor assessment was performed after randomisation, data were censored at the date of randomisation +1 day.
Time Frame: Time from randomization to the first occurrence of PD or death (Up to 68 months)
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 192 | 188
months | 3.58 [3.06 to 3.81] | 3.71 [2.83 to 4.01]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.7317, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.78 to 1.19]

9. Secondary Outcome: Objective Response Rate (ORR) in Response-evaluable Population, Subset of PD-L1-positive Population
Description: ORR was defined as percentage of participants with measurable disease at baseline who achieved a documented unconfirmed objective response (OR). OR was defined as either a complete response (CR) or a partial response (PR), as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD, in the absence of CR. Percentages have been rounded off to nearest whole number.
Time Frame: Baseline up to end of study (Up to 68 months)
Population: PD-L1 positive population included all participants randomized in the study whose PD-L1 status was tumor-infiltrating IC of 1% or greater (IC1/2/3) at the time of randomization, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. Response-evaluable Population included participants randomized in the study with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 159 | 154
percentage of participants | 28.3 [21.45 to 35.98] | 39.6 [31.83 to 47.80]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.0337, Cochran-Mantel-Haenszel; Difference in ORR = 11.31, 95% CI 2-sided [0.24 to 22.37]

10. Secondary Outcome: ORR in Response-evaluable Population, Subset of mITT Population
Description: ORR was defined as percentage of participants with measurable disease at baseline who achieved a documented unconfirmed OR. OR was defined as either a CR or PR, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR. Percentages have been rounded off to nearest whole number.
Time Frame: Baseline up to end of study (Up to 68 months)
Population: mITT population included all participants randomized under the protocol versions prior to version 4.0 (referred to as all-comers, i.e., PD-L1 (SP142)-positive and PD-L1 (SP142)-negative participants), grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. Response-evaluable Population included participants randomized in the study with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 168 | 171
percentage of participants | 32.1 [25.16 to 39.77] | 31.0 [24.16 to 38.51]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.9755, Cochran-Mantel-Haenszel; Difference in ORR = -1.15, 95% CI 2-sided [-11.63 to 9.34]

11. Secondary Outcome: Duration of Objective Response (DoR) in DoR-evaluable Population Subset of PD-L1-positive Population
Description: DoR was defined as the time from the first occurrence of a documented unconfirmed response (CR or PR) until the date of PD as determined by the investigator from tumor assessments using RECIST v1.1 or death from any cause, whichever occurs first. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: Time from the first occurrence of a documented OR until the date of PD/death (Up to 68 months)
Population: PD-L1 positive population included all participants randomized in the study whose PD-L1 status was tumor-infiltrating IC of 1% or greater (IC1/2/3) at the time of randomization, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. DOR-evaluable population included participants randomized in the study with measurable disease at baseline and an OR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 45 | 61
months | 4.14 [3.45 to 5.78] | 6.60 [4.63 to 8.02]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.1359, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.48 to 1.11]

12. Secondary Outcome: DoR in DoR-evaluable Population Subset of mITT Population
Description: as for outcome 11
Time Frame: Time from the first occurrence of a documented OR until the date of PD/death (Up to 68 months)
Population: mITT population included all participants randomized under the protocol versions prior to version 4.0 (referred to as all-comers, i.e., PD-L1(SP142)-positive and PD-L1(SP142)-negative participants), grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. DOR-evaluable population included participants randomized in the study with measurable disease at baseline and an OR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 54 | 53
months | 5.22 [3.81 to 6.60] | 5.70 [4.17 to 7.92]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.8225, Log Rank; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.63 to 1.43]

13. Secondary Outcome: Clinical Benefit Rate (CBR) in Response-evaluable Population Subset of PD-L1-positive Population
Description: CBR was defined as the percentage of participants with either an unconfirmed CR or PR or stable disease (SD) that lasts at least 6 months as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Percentages have been rounded off to nearest whole number.
Time Frame: Up to 68 months
Population: PD-L1 positive population included all participants randomized in the study whose PD-L1 status was tumor-infiltrating immune cells IC of 1% or greater (IC1/2/3) at the time of randomization, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. Response-evaluable population included participants randomized in the study with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 159 | 154
percentage of participants | 34.6 [27.23 to 42.53] | 42.9 [34.92 to 51.07]

14. Secondary Outcome: CBR in Response-evaluable Population Subset of mITT Population
Description: CBR was defined as the percentage of participants with either an unconfirmed CR or PR or SD that lasts at least 6 months as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Percentages have been rounded off to nearest whole number.
Time Frame: Up to 68 months
Population: mITT population included all participants randomized under the protocol versions prior to version 4.0 (referred to as all-comers, i.e., PD-L1(SP142)-positive and PD-L1(SP142)-negative participants), grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. Response-evaluable population included participants randomized in the study with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 168 | 171
percentage of participants | 36.3 [29.04 to 44.07] | 35.1 [27.96 to 42.74]

15. Secondary Outcome: Confirmed Objective Response Rate (C-ORR) in Response-evaluable Population Subset of PD-L1-positive Population
Description: C-ORR was defined as percentage of participants with measurable disease at baseline who achieved a documented confirmed OR. OR was defined as either a CR or PR, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR. Percentages have been rounded off to nearest whole number.
Time Frame: Up to 68 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 159 | 154
percentage of participants | 19.5 [13.65 to 26.52] | 31.2 [23.96 to 39.12]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.0172, Cochran-Mantel-Haenszel; Difference in ORR = 11.67, 95% CI 2-sided [1.47 to 21.87]

16. Secondary Outcome: C-ORR in Response-evaluable Population Subset of mITT Population
Description: as for outcome 15
Time Frame: Up to 68 months
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 168 | 171
percentage of participants | 23.2 [17.06 to 30.34] | 23.4 [17.27 to 30.46]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Stratified Analysis; Test type: Superiority; p = 0.8679, Cochran-Mantel-Haenszel; Difference in ORR = 0.18, 95% CI 2-sided [-9.41 to 9.77]

17. Secondary Outcome: DoR for Confirmed Responders (C-DoR) in C-DoR-evaluable Population Subset of PD-L1-positive Population
Description: C-DoR was defined as the time from the first occurrence of a documented confirmed response (CR or PR) until the date of PD as determined by the investigator from tumor assessments using RECIST v1.1 or death from any cause, whichever occurs first. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: Time from the first occurrence of a documented OR until the date of PD/death (Up to 68 months)
Population: PD-L1 population included all participants randomized in the study whose PD-L1 status was tumor-infiltrating IC of 1% or greater (IC1/2/3) at the time of randomization, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. C-DOR-evaluable population included participants randomized in the study with measurable disease at baseline and a confirmed OR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 31 | 48
months | 5.78 [4.21 to 8.48] | 7.92 [6.60 to 12.78]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.2846, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.46 to 1.26]

18. Secondary Outcome: C-DoR in C-DoR-evaluable Population Subset of mITT Population
Description: as for outcome 17
Time Frame: Time from the first occurrence of a documented OR until the date of PD/death (Up to 68 months)
Population: mITT population included all participants randomized under the protocol versions prior to version 4.0 (referred to as all-comers, i.e., PD-L1(SP142)-positive and PD-L1(SP142)-negative participants), grouped according to their assigned treatment arm, whether or not the assigned study treatment was received. C-DOR-evaluable population included participants randomized in the study with measurable disease at baseline and a confirmed OR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 39 | 40
months | 6.51 [4.83 to 8.48] | 7.43 [5.55 to 12.98]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Test type: Superiority; p = 0.9853, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.61 to 1.61]

19. Secondary Outcome: Time to Confirmed Deterioration (TTD) in Global Health Status/Quality of Life (GHS/QoL) According to the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) in PD-L1-positive Population
Description: TTD in GHS/QoL, defined by a minimally important decrease of ≥10 points at 2 consecutive assessment time-points on the GHS/QoL scale (Items 29, 30) of EORTC QLQ-C30, which consists of 30 questions that assess 5 aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, & six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Participant responses to questions regarding GHS (Question 29: GHS; "How would you rate your overall health during the past week?") & QoL (Question 30: QoL; "How would you rate your overall quality of life during the past week?") were assessed & were scored on a 7-point scale (1= Very poor; 7=Excellent). Scores are linearly transformed on a scale of 0 to 100, with a high score indicating better QoL.
Time Frame: Up to 68 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 177 | 177
months | 6.77 [4.30 to 32.69] | 9.43 [6.01 to NA] — The upper limit of the 95% CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Stratified Analysis; Test type: Superiority; p = 0.4117, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.63 to 1.21]

20. Secondary Outcome: TTD in GHS/QoL According to EORTC QLQ-C30 in mITT Population
Description: as for outcome 19
Time Frame: Up to 68 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 192 | 188
months | 7.66 [4.34 to 32.69] | 8.90 [5.88 to 16.82]
Statistical Analysis 1: Comparison: Placebo + Chemotherapy vs Atezolizumab + Chemotherapy; Stratified Analysis; Test type: Superiority; p = 0.7215, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.68 to 1.30]

21. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions that worsen during a study are also considered AEs.
Time Frame: From treatment initiation up to 90 days after last dose (up to 71 months)
Population: Safety-evaluable population included participants who received any amount of any study drug (atezolizumab/placebo or chemotherapy).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 294 | 293
Participants | 283 | 281

22. Secondary Outcome: Serum Concentration of Atezolizumab
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 3 and 4; Post-dose on Day 1 of Cycles 1 and 3 and Treatment Discontinuation Visit (up to 69 months) (1 Cycle= 3 weeks)
Population: Pharmacokinetic (PK)-evaluable population included participants who received any dose of study medication and who had at least one evaluable post-baseline PK sample. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/millilitre (µg/mL)
Arm/Group | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 268
micrograms/millilitre (µg/mL)
  Cycle 1 Day 1 Predose | NA (NA) — Geometric mean & geometric coefficient of variation were not estimable as samples were below the limit of quantification (BLQ).
  Cycle 1 Day 1 Post-dose: number analyzed (Participants) | 263
  Cycle 1 Day 1 Post-dose | 442 (59.7)
  Cycle 2 Day 1 Pre-dose: number analyzed (Participants) | 262
  Cycle 2 Day 1 Pre-dose | 87.2 (72.7)
  Cycle 3 Day 1 Predose: number analyzed (Participants) | 223
  Cycle 3 Day 1 Predose | 140 (42.9)
  Cycle 3 Day 1 Postdose: number analyzed (Participants) | 205
  Cycle 3 Day 1 Postdose | 517 (47.7)
  Cycle 4 Day 1 Predose: number analyzed (Participants) | 167
  Cycle 4 Day 1 Predose | 157 (104.9)
  Treatment Discontinuation: number analyzed (Participants) | 187
  Treatment Discontinuation | 120 (189.7)

23. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: Number of ADA-positive participants after drug administration was determined for participants exposed to atezolizumab. For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the baseline titer result. The sum of participants who were ADA-positive at postbaseline visits of Cycles 1 to 4 and treatment discontinuation has been reported here.
Time Frame: Cycles 1 to 4 and Treatment Discontinuation visit (up to 69 months)
Population: Safety-evaluable population included participants who received any amount of any study drug (atezolizumab/placebo or chemotherapy). Overall number analyzed included participants with data available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 275
Participants | 20

24. Secondary Outcome: Number of Participants With PD-L1 Protein Expression in Screening Tumour Tissue and Post-baseline Assessment
Time Frame: Baseline up to 68 months
Population: FAS population included all participants randomized in the study, grouped according to their assigned treatment arm, whether or not the assigned study treatment was received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 298 | 297
Participants
  Baseline IC0- Post-baseline IC 0 | 3 | 0
  Baseline IC1/2/3- Post-baseline IC 0 | 0 | 0
  Baseline IC0- Post-baseline IC1/2/3 | 0 | 0
  Baseline IC1/2/3- Post-baseline IC1/2/3 | 6 | 2

25. Other Pre Specified Outcome: OS in China Population
Description: OS was defined as time from randomization to death from any cause.
Time Frame: Time from randomization to death (Up to 68 months)
Population: As pre-specified in the SAP, analysis for China population was to be conducted based on data maturity and the estimated treatment effect from the global population. As the results for global population did not meet pre-specified criteria, a separate analysis for China subpopulation was not conducted.
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

26. Other Pre Specified Outcome: 12-month Survival Rate in China Population
Description: 12-month survival rate was defined as the percentage of participants alive 12 months after randomization.
Time Frame: 12 months
Population: As pre-specified in the SAP, analysis for China population was to be conducted based on data maturity and estimated treatment effect from the global population. As the results for global population did not meet pre-specified criteria, a separate analysis for China subpopulation was not conducted.
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

27. Other Pre Specified Outcome: 18-month Survival Rate in China Population
Description: 18-month survival rate was defined as the percentage of participants alive 18 months after randomization.
Time Frame: 18 months
Population: As pre-specified in the SAP, analysis for China population was to be conducted based on data maturity and estimated treatment effect from the global population. As the results for the global population did not meet pre-specified criteria, a separate analysis for China subpopulation was not conducted.
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

28. Other Pre Specified Outcome: PFS in China Population
Description: PFS was defined as the time from randomization to the first occurrence of PD, as determined by the investigator according to RECIST 1.1, or death from any cause, whichever occurs first.
Time Frame: Time from randomization to the first occurrence of PD or death (Up to 68 months)
Population: as for outcome 27
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

29. Other Pre Specified Outcome: ORR in China Population
Description: ORR was defined as percentage of participants with measurable disease at baseline who achieved a documented unconfirmed OR. OR was defined as either a CR or PR, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR.
Time Frame: Baseline up to end of study (Up to 68 months)
Population: As pre-specified in the SAP, analysis for China population was to be conducted based on data maturity and estimated treatment effect from the global population. As the results for the global population were did not meet pre-specified criteria, a separate analysis for China subpopulation was not conducted.
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

30. Other Pre Specified Outcome: DoR in China Population
Description: as for outcome 11
Time Frame: Time from the first occurrence of a documented OR until the date of PD/death (Up to 68 months)
Population: as for outcome 29
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

31. Other Pre Specified Outcome: CBR in China Population
Description: CBR was defined as the percentage of participants with either an unconfirmed CR or PR or SD that lasts at least 6 months as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm.
Time Frame: Up to 68 months
Population: as for outcome 29
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

32. Other Pre Specified Outcome: C-ORR in China Population
Description: C-ORR was defined as percentage of participants with measurable disease at baseline who achieved a documented confirmed OR. OR was defined as either a CR or PR, as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes must have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD, in the absence of CR.
Time Frame: Up to 68 months
Population: as for outcome 29
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

33. Other Pre Specified Outcome: C-DoR in China Population
Description: as for outcome 17
Time Frame: Time from the first occurrence of a documented OR until the date of PD/death (Up to 68 months)
Population: as for outcome 27
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

34. Other Pre Specified Outcome: TTD in GHS/QoL According to EORTC QLQ-C30 in China Population
Description: as for outcome 19
Time Frame: Up to 68 months
Population: as for outcome 27
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From treatment initiation up to 90 days after the last dose (up to 71 months)
Description: Safety-evaluable population included participants who received any amount of any study drug (atezolizumab/placebo or chemotherapy).
Arm/Group | Placebo + Chemotherapy | Atezolizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 233/294 | 226/293
Serious Adverse Events (participants affected / at risk) | 57/294 | 69/293
Other Adverse Events (participants affected / at risk) | 278/294 | 276/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Chemotherapy (N=294) | Atezolizumab + Chemotherapy (N=293)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (10) | 6 (6)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acinetobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 4 (4)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 1 (1) | 1 (1)
Mastitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (4)
Platelet count decreased (Investigations) | 7 (9) | 7 (11)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Device extrusion (Product Issues) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Chemotherapy (N=294) | Atezolizumab + Chemotherapy (N=293)
Anaemia (Blood and lymphatic system disorders) | 138 (210) | 133 (199)
Leukopenia (Blood and lymphatic system disorders) | 42 (130) | 52 (153)
Lymphopenia (Blood and lymphatic system disorders) | 17 (34) | 26 (40)
Neutropenia (Blood and lymphatic system disorders) | 119 (322) | 108 (341)
Thrombocytopenia (Blood and lymphatic system disorders) | 54 (123) | 52 (117)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 15 (17)
Hypothyroidism (Endocrine disorders) | 12 (13) | 25 (29)
Abdominal pain (Gastrointestinal disorders) | 18 (23) | 14 (16)
Abdominal pain upper (Gastrointestinal disorders) | 19 (24) | 17 (19)
Constipation (Gastrointestinal disorders) | 61 (77) | 61 (87)
Diarrhoea (Gastrointestinal disorders) | 40 (55) | 46 (75)
Dyspepsia (Gastrointestinal disorders) | 16 (19) | 8 (8)
Nausea (Gastrointestinal disorders) | 122 (179) | 121 (236)
Vomiting (Gastrointestinal disorders) | 69 (90) | 67 (109)
Asthenia (General disorders) | 73 (93) | 66 (95)
Fatigue (General disorders) | 62 (75) | 69 (85)
Mucosal inflammation (General disorders) | 14 (19) | 16 (18)
Oedema peripheral (General disorders) | 13 (14) | 17 (22)
Pyrexia (General disorders) | 39 (61) | 49 (68)
Upper respiratory tract infection (Infections and infestations) | 13 (20) | 18 (26)
Urinary tract infection (Infections and infestations) | 9 (9) | 16 (22)
Alanine aminotransferase increased (Investigations) | 100 (187) | 95 (160)
Aspartate aminotransferase increased (Investigations) | 91 (195) | 86 (138)
Blood alkaline phosphatase increased (Investigations) | 19 (26) | 19 (22)
Lymphocyte count decreased (Investigations) | 36 (60) | 23 (44)
Neutrophil count decreased (Investigations) | 88 (249) | 77 (311)
Platelet count decreased (Investigations) | 69 (171) | 69 (169)
White blood cell count decreased (Investigations) | 64 (178) | 58 (227)
Decreased appetite (Metabolism and nutrition disorders) | 32 (33) | 50 (51)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (35) | 40 (46)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (35) | 28 (30)
Bone pain (Musculoskeletal and connective tissue disorders) | 16 (22) | 10 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (20) | 19 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (30) | 24 (26)
Dizziness (Nervous system disorders) | 17 (18) | 23 (25)
Headache (Nervous system disorders) | 54 (73) | 52 (70)
Insomnia (Psychiatric disorders) | 19 (21) | 25 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (43) | 38 (44)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 19 (21)
Alopecia (Skin and subcutaneous tissue disorders) | 29 (30) | 21 (22)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 29 (34) | 32 (40)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (15) | 24 (35)
Rash (Skin and subcutaneous tissue disorders) | 22 (25) | 33 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT03371017/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03371017/SAP_001.pdf